CLINICAL TRIAL: NCT03752866
Title: CONtrolled Delivery For ImproveD outcomEs With cliNiCal Evidence
Brief Title: CONFIDENCE Registry to Assess Safety and Performance of Portico System to Treat Patients With Severe Aortic Stenosis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SJM-CIP-CL1003491
Record Dates: First submitted 2018-11-15; First posted 2018-11-26 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Symptomatic Degenerative Aortic Stenosis; Severe Aortic Stenosis
Keywords: Portico™ valve; Portico™ valve delivery system; Portico™ valve loading system; Transcatheter Aortic Valve Replacement; Aortic Stenosis; Heart Valve Prosthesis; TAVR; TAVR Registry; Transcatheter Aortic Valve Implant; TAVI; TAVI Registry; FlexNav delivery system; FlexNav loading system
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: This registry will include market released Portico™ valves (23mm, 25mm, 27mm and 29mm), delivery systems and loading systems. The registry will also allow future iterations of the Portico valve and delivery system along with expanded indications to be included as they receive approval for commercial use in the country where the subject is enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Portico™ Valve, Delivery System(s) and Loading System(s) (Experimental): Subjects undergoing implantation of a commercially available Portico transcatheter aortic heart valve using the Portico TAVI system will be included.
  Interventions: Device: Portico™ Valve, Portico Delivery System(s) and Loading System(s)
- Portico™ Valve, FlexNav Delivery and Loading System(s) (Experimental): Subjects undergoing implantation of a commercially available Portico transcatheter aortic heart valve using the FlexNav Delivery and Loading Systems will be included.
  Interventions: Device: Portico™ Valve, FlexNav Delivery System(s) and Loading System(s)

INTERVENTIONS:
Device: Portico™ Valve, Portico Delivery System(s) and Loading System(s) — Subjects will undergo implantation of a commercially available Portico transcatheter aortic heart valve using the Portico TAVI system.
  Arms: Portico™ Valve, Delivery System(s) and Loading System(s)
Device: Portico™ Valve, FlexNav Delivery System(s) and Loading System(s) — Subjects will undergo implantation of a commercially available Portico transcatheter aortic heart valve using the FlexNav Delivery and Loading Systems.
  Arms: Portico™ Valve, FlexNav Delivery and Loading System(s)

SUMMARY:
The purpose of this clinical investigation is to characterize the procedural safety and device performance of transfemoral implantation of the Portico™ Transcatheter Aortic Heart Valve in patients with symptomatic degenerative aortic stenosis.

DETAILED DESCRIPTION:
The CONFIDENCE registry study will be conducting as a prospective, non-randomized, observational, single-arm, multi-center study.

Approximately 1000 subjects with severe symptomatic (NYHA class ≥ II) aortic stenosis (AS), will undergo Portico™ Transcatheter Aortic Heart Valve implantation.

The subject data will be collected at baseline, index procedure, pre- discharge, 30 days and 12 months from the index procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are ≥18 years of age or legal age in host country and have been identified as a candidate for a Portico™ valve implant
2. Subjects who have been informed of the nature of the study, agree to its provisions and have provided written informed consent as approved by the Ethics Committee (EC) of the respective clinical center

Exclusion Criteria:

1. Have sepsis, including active endocarditis
2. Have any evidence of left ventricular or atrial thrombus
3. Have vascular conditions (i.e. caliber, stenosis, tortuosity, or severe calcification) that make insertion and endovascular access to the aortic valve improbable
4. Have a non-calcified aortic annulus
5. Have congenital bicuspid or unicuspid leaflet configuration
6. Are unable to tolerate antiplatelet/anticoagulant therapy
7. Are pregnant at the time of signing informed consent
8. Are currently participating in a drug or device study that may impact the registry (unless prior sponsor approval for co-enrollment is granted)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1001 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2022-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helge Möllmann, Principal Investigator — St. Johannes Hospital, Dortmund, Germany; Vinny Podichetty, Study Director — Abbott Structural Heart
Locations (28):
- Heart Care Partners- Wesley Hospital, Woolloongabba, Queensland, Australia
- AZ Middelheim, Antwerp, Belgium
- University Hospital Olomouc, Olomouc, Czechia
- Germany (11):
  - Kliniken der Friedrich-Alexander-Universitat, Erlangen, Bavaria
  - Kerckhoff-Klinik gGmbH, Bad Nauheim
  - Universitätsmedizin Berlin - Charité Campus Mitte (CCM), Berlin
  - Universitätsmedizin Berlin - Campus Benjamin Franklin (CBF), Berlin
  - St.-Johannes-Hospital, Dortmund
  - Herzzentrum Dresden GmbH Universitätsklinik, Dresden
  - Klinikum der Johann Wolfgang Goethe-Universität Frankfurt, Frankfurt
  - UKE Hamburg (Universitatsklinik Eppendorf), Hamburg
  - Städtisches Klinikum Karlsruhe gGmbH Medizinischen Klinik IV, Karlsruhe
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Charite Campus Virchow Klinikum, Mitte
- Italy (4):
  - Policlinico di Monza, Monza, Lombardy
  - Ospedale San Raffaele, Milan
  - Policlinico San Donato, San Donato Milanese
  - Ospedale San Bortolo, Vicenza
- Samodzielny Publiczny Centralny Szpital Kliniczny, Warsaw, Masovian Voivodeship, Poland
- Spain (4):
  - Hospital de la Santa Creu I Sant Pau, Barcelona, Catalonia
  - Hospital General Juan Ramon Jimenez, Huelva
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
- Kantonsspital Aarau, Aarau, Switzerland
- United Kingdom (4):
  - Royal Victoria Hospital, Belfast, Ireland
  - James Cook University Hoospital, Middlesbrough, North East England
  - Morriston Hospital - ABM University Health Board, Morriston, Swansea
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mollmann H, Linke A, Nombela-Franco L, Sluka M, Francisco Oteo Dominguez J, Montorfano M, Kim WK, Arnold M, Vasa-Nicotera M, Fichtlscherer S, Conradi L, Camuglia A, Bedogni F, Kohli K, Manoharan G. Valve Hemodynamics by Valve Size and 1-Year Survival Following Implantation of the Portico Valve in the Multicenter CONFIDENCE Registry. Struct Heart. 2023 Nov 11;8(1):100226. doi: 10.1016/j.shj.2023.100226. eCollection 2024 Jan. PMID 38283573

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 2018 and July 2021, implantation with a Portico™ transcatheter heart valve (THV) was attempted in 1001 subjects. This clinical investigation includes 27 sites in 8 countries across Europe and 1 site in Australia.
Groups:
- Portico™ Valve, Delivery System(s) and Loading System(s): Implantation of the Portico ™ Valve using the Portico Delivery and Loading Systems. Subjects will undergo implantation of a commercially available Portico transcatheter aortic heart valve using the Portico TAVI system.
- Portico™ Valve, FlexNav Delivery and Loading System(s): Implantation of the Portico ™ Valve using the FlexNav Delivery and Loading Systems. Subjects will undergo implantation of a commercially available Portico transcatheter aortic heart valve using the FlexNav Delivery and Loading Systems.
Period: Overall Study
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s)
Started | 501 | 500
Completed | 501 | 500
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s) | Total
Number analyzed (Participants) | 501 | 500 | 1001
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.7 (5.4) | 82.3 (5.3) | 82.0 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 319 | 307 | 626
  Male | 182 | 193 | 375
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 4 | 0 | 4
  Czechia | 25 | 42 | 67
  Poland | 10 | 24 | 34
  Italy | 43 | 68 | 111
  United Kingdom | 44 | 25 | 69
  Australia | 20 | 8 | 28
  Switzerland | 12 | 0 | 12
  Germany | 272 | 195 | 467
  Spain | 71 | 138 | 209
Hypertension [Count of Participants; unit: Participants] | 440 | 431 | 871
NYHA Classification [Count of Participants; unit: Participants] — New York Heart Association heart failure classification. I - no symptoms and no limitation. II - mild symptoms. III - marked limitation in activity due to symptoms, even during less-than-ordinary activity.
  IV - severe limitation, experiences symptoms even at rest.
  Participants
    NYHA I | 14 | 4 | 18
    NYHA II | 160 | 185 | 345
    NYHA III | 295 | 293 | 588
    NYHA IV | 32 | 18 | 50
Baseline EQ5D-3L Visual Analog Scale Value [Mean (Standard Deviation); unit: units on a scale] — EQ5D-3L stands for EuroQol5D-3L. Scale 0-100 (best). Subject selects their rating of their own health on a visual scale from 0-100.
  Scores were used as a measure of improvement from baseline; subjects served as their own controls. Staging was relative to the unitless baseline score - higher score was better. Population: The number analyzed in row differs because not all subjects had EQ5D-3L collected at baseline.
  units on a scale
    number analyzed (Participants) | 406 | 458 | 864
    (all) | 60.8 (18.5) | 60.1 (17.8) | 60.4 (18.1)

OUTCOME MEASURES:

1. Primary Outcome: Cardiovascular Mortality
Description: Death due to proximate cardiac cause, non-coronary vascular conditions, procedure-related deaths, valve-related deaths, sudden or unwitnessed death and unknown cause.
Time Frame: 30 days from the index procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s)
Number analyzed (Participants) | 501 | 500
Participants | 15 | 6

2. Secondary Outcome: Number of Subjects With Myocardial Infarction
Time Frame: At 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s)
Number analyzed (Participants) | 501 | 500
Participants | 2 | 1

3. Secondary Outcome: Number of Subjects With Stroke
Time Frame: At 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s)
Number analyzed (Participants) | 501 | 500
Participants
  Disabling Stroke | 8 | 10
  Non-Disabling Stroke | 5 | 6

4. Secondary Outcome: Number of Subjects With Bleeding Events
Time Frame: At 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s)
Number analyzed (Participants) | 501 | 500
Participants
  Life Threatening | 16 | 18
  Major | 26 | 33
  Minor | 31 | 20

5. Secondary Outcome: Number of Subjects With Acute Kidney Injury
Description: The increase in creatinine must occur within 48 hours.
  Stage 1: Increase in serum creatinine to 150% to 199% (1.5 to 1.99 X increase compared with baseline) or increase of greater than or equal to 0.3 mg/dL (26.4 mmol/L) or Urine output <0.5 mL/kg per hour for >6 but <12 hours.
  Stage 2: Increase in serum creatinine to 200% to 299% (2.0 to 2.99 X increase compared with baseline) or Urine output <0.5 mL/kg per hour for >12 but <24 hours.
  Stage 3: Increase in serum creatinine to greater than or equal to 300% (3 X increase compared with baseline) or serum creatinine of ≥ 4.0 mg/dL (354 mmol/L) with an acute increase of at least 0.5 mg/dL (44 mmol/L)or Urine output <0.3 mL/kg per hour for ≥24 hours or anuria for ≥12 hours. Patients receiving renal replacement therapy are considered to meet Stage 3 criteria irrespective of other criteria.
Time Frame: At 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s)
Number analyzed (Participants) | 501 | 500
Participants
  Stage 1 | 4 | 5
  Stage 2 | 0 | 3
  Stage 3 | 7 | 4

6. Secondary Outcome: Number of Subjects With Vascular Complications
Time Frame: At 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s)
Number analyzed (Participants) | 501 | 500
Participants
  Major | 32 | 41
  Minor | 36 | 25

7. Secondary Outcome: Number of Subjects With Annular Rupture
Time Frame: At 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s)
Number analyzed (Participants) | 501 | 500
Participants | 2 | 1

8. Secondary Outcome: Number of Subjects With Coronary Obstruction
Time Frame: At 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s)
Number analyzed (Participants) | 501 | 500
Participants | 2 | 3

9. Secondary Outcome: Number of Subjects Undergoing Conversion To Open Surgery
Time Frame: At 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s)
Number analyzed (Participants) | 501 | 500
Participants | 3 | 3

10. Secondary Outcome: Number Of Subjects Undergoing Transcatheter Valve-In-Valve Deployment
Time Frame: At 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s)
Number analyzed (Participants) | 501 | 500
Participants | 3 | 6

11. Secondary Outcome: Number Of Subjects With Valve Embolization
Time Frame: At 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s)
Number analyzed (Participants) | 501 | 500
Participants | 6 | 7

12. Secondary Outcome: Number Of Subjects Undergoing Naïve Permanent Pacemaker Insertion
Time Frame: At 30 days
Population: Subjects with a pacemaker at baseline are not included.
Measure: Count of Participants; unit: Participants
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s)
Number analyzed (Participants) | 454 | 444
Participants | 87 | 84

13. Secondary Outcome: Vessel Diameter
Time Frame: At 30 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s)
Number analyzed (Participants) | 499 | 497
mm | 7.42 (1.44) | 7.09 (1.36)

14. Secondary Outcome: Introducer Sheath Used
Description: This is a yes or no question on the CRF. Sites report if the implanter used an introducer sheath (a special device used to facilitate introduction of the investigational device into the subjects vasculature).
Time Frame: At 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s)
Number analyzed (Participants) | 501 | 500
Participants | 469 | 120

15. Secondary Outcome: Implant Success
Time Frame: At 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s)
Number analyzed (Participants) | 501 | 500
Participants | 488 | 488

16. Secondary Outcome: Effective Orifice Area
Description: Effective orifice area is a measure of the working area of the implanted valve determined by echocardiograph.
Time Frame: At 30 days
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s)
Number analyzed (Participants) | 320 | 283
cm^2 | 1.85 (0.48) | 1.80 (0.49)

17. Secondary Outcome: Aortic Valve Mean Gradient
Description: Aortic valve mean gradient is a measure of the pressure gradient across the aortic valve measured by echocardiograph.
Time Frame: At 30 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s)
Number analyzed (Participants) | 404 | 405
mmHg | 7.38 (4.44) | 6.80 (2.79)

18. Secondary Outcome: Number of Subjects With Paravalvular Leak (PVL)
Time Frame: At 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s)
Number analyzed (Participants) | 382 | 386
Participants
  None/Trace/Trivial | 185 | 158
  Mild | 188 | 221
  Moderate | 9 | 7
  Severe | 0 | 0

19. Secondary Outcome: NYHA Classification
Description: NYHA Functional Classification is a system used to assess patient heart failure severity based on their limitations of physical activity. The four classes are described below:
  Class I: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, or shortness of breath.
  Class II: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath or chest pain.
  Class III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain.
  Class IV: Symptoms of heart failure at rest. Any physical activity causes further discomfort.
  Subjects' NYHA Classification based on above criteria was assessed during follow up, and subjects were assigned to one of four classifications. Results are presented as percentage of all available subjects who were assigned each functional class (I-IV).
Time Frame: At 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s)
Number analyzed (Participants) | 431 | 457
Participants
  NYHA I | 152 | 159
  NYHA II | 218 | 254
  NYHA III | 58 | 42
  NYHA IV | 3 | 2

20. Secondary Outcome: EQ5D-3L Visual Analog Scale Value
Description: The EQ-5D-3L consists of EuroQoL 5 questions and 3 answering levels. The rating of questions includes: Level 1 no problems; Level 2 some problems; Level 3 Significant problems; Worst case is 15 points; and best case is 5 points using index. The Visual analogue scale VAS 0-100 where 0 is the worst imaginable health state and 100 the best imaginable health state."
Time Frame: At 30 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s)
Number analyzed (Participants) | 406 | 458
units on a scale | 66.5 (18.3) | 66.0 (18.0)

21. Secondary Outcome: Kaplan-Meier Rate of All-cause Mortality
Description: Kaplan-Meier (KM) percentage of subjects who died. KM is a statistical method that attempts to account for other factors that may have reduced the number of subjects evaluable at a given time point.
Time Frame: At 12 months
Measure: Number; unit: percentage of All-cause Mortality
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s)
Number analyzed (Participants) | 501 | 500
percentage of All-cause Mortality | 13.7 | 11.0

ADVERSE EVENTS:
Time Frame: 30 days
Description: The adverse event data were collected for 30 days. However, the all-Cause mortality was assessed for up to 12 months.
Arm/Group | Portico™ Valve, Delivery System(s) and Loading System(s) | Portico™ Valve, FlexNav Delivery and Loading System(s)
All-Cause Mortality (participants affected / at risk) | 16/501 | 10/500
Serious Adverse Events (participants affected / at risk) | 348/501 | 358/500
Other Adverse Events (participants affected / at risk) | 72/501 | 80/500
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Portico™ Valve, Delivery System(s) and Loading System(s) (N=501) | Portico™ Valve, FlexNav Delivery and Loading System(s) (N=500)
Anemia (Blood and lymphatic system disorders) | 12 | 12
Other (Blood and lymphatic system disorders) | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 5
Thrombus (Blood and lymphatic system disorders) | 1 | 0
Aortic Valve Regurgitation (Cardiac disorders) | 1 | 3
Atrial Fibrillation (Cardiac disorders) | 7 | 12
Atrial Flutter (Cardiac disorders) | 1 | 1
Bleeding (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 4 | 4
Cardiac Arrhythmias (Cardiac disorders) | 6 | 9
Cardiogenic Shock (Cardiac disorders) | 4 | 0
Complete Heart Block (Cardiac disorders) | 59 | 49
Congestive Heart Failure (Cardiac disorders) | 10 | 15
Death - Unknown (Cardiac disorders) | 18 | 16
Dyspnea (Cardiac disorders) | 2 | 3
Endocarditis (Cardiac disorders) | 4 | 2
First Degree Heart Block (Cardiac disorders) | 3 | 2
Hypertension (Cardiac disorders) | 0 | 1
Hypotension (Cardiac disorders) | 0 | 1
Left Bundle Branch Block (Cardiac disorders) | 13 | 9
Mitral Valve Insufficiency (Cardiac disorders) | 1 | 3
Myocardial Infarction (Cardiac disorders) | 2 | 4
Myocardial Ischemia (Cardiac disorders) | 2 | 0
Other (Cardiac disorders) | 34 | 32
Paravalvular Leak (Cardiac disorders) | 5 | 2
Pericardial Effusion (Cardiac disorders) | 0 | 3
Pericardial Tamponade (Cardiac disorders) | 2 | 3
Pleural Effusion (Cardiac disorders) | 0 | 1
Respiratory Failure (Cardiac disorders) | 0 | 1
Second Degree Heart Block (Cardiac disorders) | 1 | 2
Thrombus On Device (Cardiac disorders) | 0 | 1
Valve Embolization (Cardiac disorders) | 0 | 1
Ventricular Fibrillation (Cardiac disorders) | 2 | 0
Ventricular Tachycardia (Cardiac disorders) | 0 | 1
Other (Endocrine disorders) | 1 | 1
Anemia (Gastrointestinal disorders) | 0 | 1
GI Bleed (Gastrointestinal disorders) | 0 | 2
Ischemia (Gastrointestinal disorders) | 2 | 0
Other (Gastrointestinal disorders) | 3 | 3
Weakness (Gastrointestinal disorders) | 0 | 1
Death - Unknown (General disorders) | 1 | 3
Fever (General disorders) | 0 | 1
Multi Organ Failure (General disorders) | 1 | 0
Other (General disorders) | 3 | 2
Other (Hepatobiliary disorders) | 3 | 0
Death - Unknown (Infections and infestations) | 0 | 2
Dyspnea (Infections and infestations) | 1 | 0
Fever (Infections and infestations) | 2 | 0
Infection (Infections and infestations) | 11 | 21
Multi Organ Failure (Infections and infestations) | 2 | 1
Other (Infections and infestations) | 10 | 9
Renal Insufficiency/Worsening Renal Function (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 5 | 4
Urinary Tract Infection/UTI (Infections and infestations) | 2 | 3
Annulus Rupture (Injury, poisoning and procedural complications) | 2 | 0
Valve Embolization (Injury, poisoning and procedural complications) | 0 | 3
Valve Migration (Injury, poisoning and procedural complications) | 2 | 3
Other (Metabolism and nutrition disorders) | 0 | 1
Other (Musculoskeletal and connective tissue disorders) | 1 | 2
Death - Unknown (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Death - Unknown (Nervous system disorders) | 0 | 2
Other (Nervous system disorders) | 6 | 8
Stroke (Nervous system disorders) | 14 | 16
Transient Ischemic Attack (TIA) (Nervous system disorders) | 2 | 1
Other (Psychiatric disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 5 | 5
Multi Organ Failure (Renal and urinary disorders) | 1 | 0
Other (Renal and urinary disorders) | 5 | 1
Renal Failure (Renal and urinary disorders) | 1 | 5
Renal Insufficiency/Worsening Renal Function (Renal and urinary disorders) | 6 | 3
Other (Reproductive system and breast disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Other (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Other (Skin and subcutaneous tissue disorders) | 1 | 2
Other (Surgical and medical procedures) | 0 | 1
Access Site Bleeding Event (Vascular disorders) | 4 | 8
Bleeding (Vascular disorders) | 14 | 12
Death - Unknown (Vascular disorders) | 1 | 0
Hematoma (Vascular disorders) | 4 | 2
Hemorrhage (Vascular disorders) | 0 | 3
Ischemia (Vascular disorders) | 1 | 1
Other (Vascular disorders) | 8 | 4
Pseudoaneurysm (Vascular disorders) | 3 | 4
Vascular Access Site And Access Related Complications (Vascular disorders) | 4 | 6
Vascular Perforation (Vascular disorders) | 4 | 1
Vascular Stenosis (Vascular disorders) | 2 | 1
Vessel Occlusion (Vascular disorders) | 4 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Portico™ Valve, Delivery System(s) and Loading System(s) (N=501) | Portico™ Valve, FlexNav Delivery and Loading System(s) (N=500)
Left Bundle Branch Block (Cardiac disorders) | 72 | 80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/66/NCT03752866/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT03752866/SAP_001.pdf